CLINICAL TRIAL: NCT04147260
Title: Partially-blind, Randomized, Parallel Group, Placebo and Active Comparator-controlled Phase I Clinical Trial to Evaluate the Photosensitivity Potential of BI 730357
Brief Title: Evaluation of Photosafety of BI 730357 Compared to Placebo and the Known Photosensitizing Agent Ciprofloxacin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1407-0037
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2022-08

CONDITIONS: Healthy
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 730357 low dose (Experimental)
  Interventions: Drug: BI 730357
- Ciprofloxacin (Active Comparator)
  Interventions: Drug: Ciprofloxacin
- BI 730357 high dose (Experimental)
  Interventions: Drug: BI 730357
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo to match BI 730357

INTERVENTIONS:
Drug: BI 730357 — Film-coated tablet
  Arms: BI 730357 high dose; BI 730357 low dose
Drug: Placebo to match BI 730357 — Film-coated tablet
  Arms: Placebo
Drug: Ciprofloxacin — Film-coated tablet
  Arms: Ciprofloxacin

SUMMARY:
To evaluate the photosensitivity potential of BI 730357

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects according to the assessment of the Investigator, based on a complete medical history, physical examination (including dermatological skin type assessment), vital signs (blood pressure, pulse rate), 12-lead ECG, and clinical laboratory tests
* 18 to 55 years old
* BMI 18 to 35 kg/m (incl.)
* Fitzpatrick skin type I, II, or III:

  * I Always burns easily, never tans
  * II Always burns easily, tans minimally
  * III Burns moderately, tans gradually
* No ultraviolet exposure of the test areas 4 weeks prior to baseline photo testing
* Normal skin response during preliminary photo testing.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
* Women of childbearing potential (WOCBP)1 must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information

Exclusion Criteria:

* Any finding in the medical examination (including blood pressure, pulse rate or ECG) deviating from normal and judged as clinically relevant by the Investigator.
* Any laboratory value outside the reference range that the Investigator considers to be of clinical relevance.
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders or any evidence of a concomitant disease judged as clinically relevant by the Investigator.
* Major surgery (major according to the investigator's assessment) performed within 10 weeks prior to randomisation or planned within 2 months after screening.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Active skin disorders on the back where photosensitivity testing will be performed.
* Subjects who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Subjects not expected to comply with the protocol requirements or not expected to complete the trial as scheduled (e.g. chronic alcohol or drug abuse or any other condition that, in the investigator's opinion, makes the subject an unreliable trial participant).
* Currently enrolled in another investigational device or drug trial, or less than 30 days (or 5 half-lives (whichever longer)) since ending another investigational drug trial.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients).
* History of hypersensitivity to ciprofloxacin, any member of the quinolone class of antibacterials.
* History of hypersensitivity to sunlight or artificial source of intense light, especially UV light.
* Chronic or acute infections which are of relevance in the opinion of the Investigator.
* Positive result for HIV, HBV, and hepatitis C (Hep C) at screening.
* History of TB or positive finding in IGRA.
* Unwillingness/inability to refrain from intake of alcoholic beverages from 48 hours prior to the trial medication administration and until Day 7 post trial medication administration.
* Positive drug screening.
* Blood donation of more than 500 mL within 30 days prior to administration of trial medication or intended donation during the trial.
* Intention to perform excessive physical activities within 4 days prior to administration of trial medication or contact sport during the entire trial and unwilling to avoid vigorous exercise for 7 days post dosing.
* Inability to comply with dietary regimen of trial site.
* Unwillingness to adhere to the rules of UV-light protection
* Received a live vaccination within 12 weeks prior to randomisation (visit 2), or any plan to receive a live vaccination during the conduct of this trial.
* Subjects with known prolongation of the QT interval, risk factors for QT prolongation or torsade de pointes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research, Inc., Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a partially blind, randomized, parallel group, placebo, and active comparator controlled Phase I clinical trial in healthy male and female subjects to evaluate the photosensitivity potential of BI 730357 compared with placebo and active comparator, and to assess the relationship between the photosensitivity response and pharmacokinetics of BI 730357.
Pre-assignment Details: All subjects were screened for eligibility to participants in the trial. Subjects attended specialist sites which would then ensure that they met all strictly implemented inclusion/exclusion criteria. Subjects were not to be assigned to treatment groups if any one of the specific entry criteria were violated.
Groups:
- Placebo QD: Subjects received orally, four Placebo film-coated tablets once per day (QD) over 8 days. Medication administration was to take place at the same time every day within a deviation of no more than ±15 minutes together with about 240 millilitres (mL) of water.
- 400 mg QD BI 730357: Subjects received orally, four BI 730357 film-coated tablets of 100 miligrams (mg) each (400 mg in total) once per day (QD) over 8 days. Medication administration was to take place at the same time every day within a deviation of no more than ±15 minutes together with about 240 mL of water.
- Placebo BID: Subjects received orally, three Placebo film-coated tablets two times per day (BID) over 7 days with a single dose Placebo on Day 8. Medication administration was to take place at the same time every day within a deviation of no more than ±15 minutes together with about 240 mL of water.
- 300 mg BID BI 730357: Subjects received orally, three BI 730357 film-coated tablets of 100 miligrams (mg) each, two times per day (BID) (2 x 300 mg = 600 mg daily dose in total) over 7 days with a single dose of 300 mg on Day 8. Medication administration was to take place at the same time every day within a deviation of no more than ±15 minutes together with about 240 mL of water.
- 500 mg Ciprofloxacin (Active Comparator): Subjects received orally, one Ciprofloxacin film-coated tablet of 500 miligrams (mg) each, two times per days (BID) (2 x 500 mg = 1000 mg daily dose in total) over 5 days from day 3 with a single dose of 500 mg on Day 8. Medication administration was to take place at the same time every day within a deviation of no more than ±15 minutes together with about 240 mL of water.
Period: Overall Study
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Started | 9 | 27 | 9 | 28 | 12
Completed | 8 | 27 | 7 | 25 | 12
Not Completed | 1 | 0 | 2 | 3 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS included all subjects who were randomized and treated with at least 1 dose of investigational product (IP) (BI 730357, placebo, or Ciprofloxacin). The TS was used for safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator) | Total
Number analyzed (Participants) | 9 | 27 | 9 | 28 | 12 | 85
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (12.06) | 37.0 (11.62) | 40.1 (8.84) | 39.7 (12.84) | 40.7 (12.58) | 39.4 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 12 | 6 | 18 | 3 | 43
  Male | 5 | 15 | 3 | 10 | 9 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 14 | 6 | 12 | 5 | 41
  Not Hispanic or Latino | 5 | 13 | 3 | 16 | 7 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Unknown or Not Reported group is actually Other
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 1 | 1 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    White | 9 | 26 | 7 | 26 | 12 | 80
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2
Minimum Erythema Dose (MED) at baseline under condition 1 [Mean (Standard Deviation); unit: millijoules/squarecentimeter] — MED defined as lowest dose that produced uniform redness (condition 1) (assessed in mJ for UVB/UVA).
  Condition 1: under full range solar UVB/UVA (290 to 400 nm, UBV content ~10%), simulating midday summer outdoor sun exposure (assessed in μw/cm2) Subjects were exposed to series of 6 graded full range solar UVB/UVA exposures, each 25% greater than previous dose. Outpatient irradiation and baseline MED testing for Irradiation Condition 1 occurred on Day -2. Two areas of back were defined for irradiation, followed by MED assessments at 24 hours (±10) minutes (Day -1) post irradiation. Population: Full Analysis Set (FAS): This set included all subjects in the treated set (TS) who provided at least 1 photosensitivity endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of photosensitivity.
  millijoules/squarecentimeter
    number analyzed (Participants) | 8 | 27 | 7 | 25 | 12 | 79
    (all) | 30.60 (6.328) | 35.41 (11.892) | 36.84 (7.910) | 30.82 (12.163) | 30.78 (12.280) | 32.89 (11.34)
Minimum Erythema Dose (MED) at baseline under condition 2 [Mean (Standard Deviation); unit: Joules/squarecentimeter] — MED = lowest dose that produced uniform darkening (condition 2 C2) (in J for UVA). C2: UVA only (320 to 400 nm, UVB content <0.03%), simulating indoor exposure behind window glass with 2. assessment of erythema + local skin reactions at 25 Joules per centimetres-2 (J cm-2) (assessed in mw/cm2) Subjects exposed to series of 6 graded full range solar UVA exposures, each 25% greater than previous dose. Outpatient irradiation and baseline MED testing for Irradiation C2 occurred Day -2. Two areas of back defined for irradiation, MED assessments at 24 hours (±10) minutes (Day -1) post irradiation. Population: Full Analysis Set (FAS): This set included all subjects in the treated set (TS) who provided at least 1 photosensitivity endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of photosensitivity.
  Joules/squarecentimeter
    number analyzed (Participants) | 8 | 27 | 7 | 25 | 12 | 79
    (all) | 21.60 (4.04) | 24.09 (2.76) | 25.10 (0.00) | 20.83 (5.29) | 22.58 (4.64) | 22.67 (4.25)

OUTCOME MEASURES:

1. Primary Outcome: Photosensitivity Index at 24 Hours Under Condition 1 (i.e., Under Full Range of UVB/UVA Exposure, Simulating Midday Summer Outdoor Sun Exposure)
Description: Photosensitivity index (PI) under condition 1 (C1)(i.e., under full range solar UVB/UVA (290 to 400 nm, UBV content ~10%), simulating midday summer outdoor sun exposure (assessed in μw/cm2)), was defined as ratio of the precise Minimum erythema dose (MED)baseline to MEDon-drug at each respective post irradiation time point (i.e. 24 hours)(i.e., MEDon-drug[millijoules (mJ)]/MEDbaseline[mJ]) and was hence unitless.
  MED was defined as lowest dose that produced uniform redness (C1) (assessed in mJ for UVB/UVA).
  Subjects were exposed to a series of 6 graded full range solar UVB/UVA exposures, each 25% greater than the previous dose.
  Light exposure occurred 2 hours (±10 minutes) after dose on Day 8 of either investigational product (IP) or placebo, and on-treatment photosensitivity assessments (determination of MEDon-drug + evaluation of erythema/local skin reactions) were performed at 24 hours after irradiation.
Time Frame: At 24 hours after irradiation on Day 8
Population: Full Analysis Set (FAS): This set included all subjects in the treated set (TS) who provided at least 1 photosensitivity endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of photosensitivity.
Measure: Least Squares Mean (95% Confidence Interval); unit: Unitless
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Number analyzed (Participants) | 8 | 27 | 7 | 25 | 12
Unitless | 0.93 [0.80 to 1.05] | 1.01 [0.95 to 1.08] | 1.00 [0.88 to 1.12] | 1.04 [0.98 to 1.11] | 1.08 [0.98 to 1.17]
Statistical Analysis 1: Comparison: Placebo QD vs 400 mg QD BI 730357; Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; Test type: Equivalence — Two-sided 90% CI with an acceptance range of -0.4 to 0.4; Linear mixed model; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.09, 90% CI 2-sided [-0.03 to 0.20], Standard Error of Mean 0.068
Statistical Analysis 2: Comparison: Placebo BID vs 300 mg BID BI 730357; Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; Test type: Equivalence — Two-sided 90% CI with an acceptance range of -0.4 to 0.4; Linear mixed model; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.04, 90% CI 2-sided [-0.07 to 0.16], Standard Error of Mean 0.067
Statistical Analysis 3: Comparison: 300 mg BID BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.572, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.03, 90% CI 2-sided [-0.14 to 0.08], Standard Error of Mean 0.055
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.315, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.08, 90% CI 2-sided [-0.07 to 0.23], Standard Error of Mean 0.075
Statistical Analysis 5: Comparison: 400 mg QD BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.286, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.06, 90% CI 2-sided [-0.18 to 0.05], Standard Error of Mean 0.059
Statistical Analysis 6: Comparison: Placebo QD vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.057, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.15, 90% CI 2-sided [0.00 to 0.31], Standard Error of Mean 0.077

2. Primary Outcome: Photosensitivity Index at 24 Hours Under Condition 2 (i.e., Under UVA Exposure Only, Simulating Indoor Sun Exposure Behind Window Glass)
Description: Photosensitivity index (PI) under condition 2 (C2)(i.e., UVA only (320 to 400 nm, UVB content <0.03%), simulating indoor exposure behind window glass with a secondary assessment of erythema and local skin reactions at 25 Joules per centimetres-2 (J cm-2) (assessed in mw/cm2)), defined as ratio of the precise Minimum erythema dose (MED)baseline to MEDon-drug at each respective post irradiation time point (i.e. 24 hours)(i.e., MEDon-drug[Joules (J)]/MEDbaseline[J]) and hence unitless.
  MED was defined as lowest dose that produced uniform darkening (C2) (assessed in J for UVA).
  Subjects were exposed to series of 6 graded full range solar UVA exposures (C2), each 25% greater than the previous dose.
  Light exposure occurred 2 hours (±10 minutes) after dose on Day 8 of either investigational product (IP) or placebo, and on-treatment photosensitivity assessments (determination of MEDon-drug + evaluation of erythema/local skin reactions) were performed at 24 hours after irradiation.
Time Frame: At 24 hours after irradiation on Day 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Unitless
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Number analyzed (Participants) | 8 | 27 | 7 | 25 | 12
Unitless | 0.94 [0.67 to 1.21] | 1.17 [1.02 to 1.32] | 1.00 [0.78 to 1.22] | 1.01 [0.89 to 1.13] | 1.52 [1.35 to 1.69]
Statistical Analysis 1: Comparison: Placebo QD vs 400 mg QD BI 730357; Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; Test type: Equivalence — Two-sided 90% CI with an acceptance range of -0.4 to 0.4; Linear mixed model; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.23, 90% CI 2-sided [-0.02 to 0.49], Standard Error of Mean 0.153
Statistical Analysis 2: Comparison: Placebo BID vs 300 mg BID BI 730357; Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; Test type: Equivalence — Two-sided 90% CI with an acceptance range of -0.4 to 0.4; Linear mixed model; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.01, 90% CI 2-sided [-0.20 to 0.22], Standard Error of Mean 0.124
Statistical Analysis 3: Comparison: 300 mg BID BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p < 0.001, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.51, 90% CI 2-sided [-0.72 to -0.31], Standard Error of Mean 0.102
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p < 0.001, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.52, 90% CI 2-sided [0.24 to 0.80], Standard Error of Mean 0.138
Statistical Analysis 5: Comparison: 400 mg QD BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.010, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.35, 90% CI 2-sided [-0.62 to -0.09], Standard Error of Mean 0.132
Statistical Analysis 6: Comparison: Placebo QD vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.001, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.59, 90% CI 2-sided [0.24 to 0.93], Standard Error of Mean 0.173

3. Secondary Outcome: Photosensitivity Index (PI) at 10 Minutes Under Condition 1 (i.e., Under Full Range of UVB/UVA Exposure, Simulating Midday Summer Outdoor Sun Exposure)
Description: Photosensitivity index (PI) under condition 1 (C1)(i.e., under full range solar UVB/UVA (290 to 400 nm, UBV content ~10%), simulating midday summer outdoor sun exposure (assessed in μw/cm2)), was defined as ratio of the precise Minimum erythema dose (MED)baseline to MEDon-drug at each respective post irradiation time point (i.e. 10 minutes)(i.e., MEDon-drug[millijoules (mJ)]/MEDbaseline[mJ]) and was hence unitless.
  MED was defined as lowest dose that produced uniform redness (C1) (assessed in mJ for UVB/UVA).
  Subjects were exposed to a series of 6 graded full range solar UVB/UVA exposures, each 25% greater than the previous dose.
  Light exposure occurred 2 hours (±10 minutes) after dose on Day 8 of either investigational product (IP) or placebo, and on-treatment photosensitivity assessments (determination of MEDon-drug + evaluation of erythema/local skin reactions) were performed at 10 minutes after irradiation.
Time Frame: At 10 minutes after irradiation on Day 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Unitless
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Number analyzed (Participants) | 8 | 27 | 7 | 25 | 12
Unitless | 0.98 [0.90 to 1.05] | 1.00 [0.96 to 1.04] | 1.00 [0.82 to 1.18] | 1.06 [0.97 to 1.16] | 1.00 [0.94 to 1.06]
Statistical Analysis 1: Comparison: Placebo QD vs 400 mg QD BI 730357; Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; Test type: Equivalence — Two-sided 90% CI with an acceptance range of -0.4 to 0.4; Linear mixed model; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.03, 90% CI 2-sided [-0.05 to 0.10], Standard Error of Mean 0.044
Statistical Analysis 2: Comparison: 400 mg QD BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.998, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.00, 90% CI 2-sided [-0.08 to 0.08], Standard Error of Mean 0.038
Statistical Analysis 3: Comparison: Placebo QD vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.618, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.02, 90% CI 2-sided [-0.08 to 0.13], Standard Error of Mean 0.050
Statistical Analysis 4: Comparison: Placebo BID vs 300 mg BID BI 730357; Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; Test type: Equivalence — Two-sided 90% CI with an acceptance range of -0.4 to 0.4; Linear mixed model; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.06, 90% CI 2-sided [-0.10 to 0.23], Standard Error of Mean 0.099
Statistical Analysis 5: Comparison: 300 mg BID BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.451, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.06, 90% CI 2-sided [-0.10 to 0.23], Standard Error of Mean 0.081
Statistical Analysis 6: Comparison: Placebo BID vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 1.000, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.00, 90% CI 2-sided [-0.22 to 0.22], Standard Error of Mean 0.110

4. Secondary Outcome: Photosensitivity Index (PI) at 10 Minutes Under Condition 2 (i.e., Under UVA Exposure Only, Simulating Indoor Sun Exposure Behind Window Glass)
Description: Photosensitivity index (PI) under condition 2 (C2)(i.e., UVA only (320 to 400 nm, UVB content <0.03%), simulating indoor exposure behind window glass with secondary assessment of erythema and local skin reactions at 25 Joules centimetres-2 (J cm-2) (assessed in mw/cm2)), was defined as ratio of precise Minimum erythema dose (MED)baseline to MEDon-drug at each respective post irradiation time point (i.e. 10 minutes)(i.e., MEDon-drug[Joules (J)]/MEDbaseline[J]) and was hence unitless.
  MED defined as lowest dose that produced uniform darkening (C2) (assessed in J for UVA).
  Subjects were exposed to series of 6 graded full range solar UVA exposures (C2), each 25% greater than the previous dose.
  Light exposure occurred 2 hours (±10 minutes) after dose on Day 8 of either investigational product (IP) or placebo, and on-treatment photosensitivity assessments (determination of MEDon-drug + evaluation of erythema/local skin reactions) were performed at 10 minutes after irradiation.
Time Frame: At 10 minutes after irradiation on Day 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Unitless
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Number analyzed (Participants) | 8 | 27 | 7 | 25 | 12
Unitless | 1.02 [0.76 to 1.29] | 1.13 [0.99 to 1.28] | 1.00 [0.67 to 1.33] | 1.29 [1.12 to 1.46] | 1.03 [0.81 to 1.25]
Statistical Analysis 1: Comparison: Placebo QD vs 400 mg QD BI 730357; Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; Test type: Equivalence — Two-sided 90% CI with an acceptance range of -0.4 to 0.4; Linear mixed model; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.11, 90% CI 2-sided [-0.15 to 0.36], Standard Error of Mean 0.152
Statistical Analysis 2: Comparison: 400 mg QD BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.446, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.10, 90% CI 2-sided [-0.16 to 0.36], Standard Error of Mean 0.131
Statistical Analysis 3: Comparison: Placebo QD vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.972, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.01, 90% CI 2-sided [-0.34 to 0.35], Standard Error of Mean 0.172
Statistical Analysis 4: Comparison: Placebo BID vs 300 mg BID BI 730357; Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; Test type: Equivalence — Two-sided 90% CI with an acceptance range of -0.4 to 0.4; Linear mixed model; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.29, 90% CI 2-sided [-0.02 to 0.60], Standard Error of Mean 0.182
Statistical Analysis 5: Comparison: 300 mg BID BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.091, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.26, 90% CI 2-sided [-0.04 to 0.56], Standard Error of Mean 0.150
Statistical Analysis 6: Comparison: Placebo BID vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.880, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.03, 90% CI 2-sided [-0.38 to 0.44], Standard Error of Mean 0.203

5. Secondary Outcome: Photosensitivity Index (PI) at 1 Hour Under Condition 1 (i.e., Under Full Range of UVB/UVA Exposure, Simulating Midday Summer Outdoor Sun Exposure)
Description: Photosensitivity index (PI) under condition 1 (C1)(i.e., under full range solar UVB/UVA (290 to 400 nm, UBV content ~10%), simulating midday summer outdoor sun exposure (assessed in μw/cm2)), was defined as ratio of the precise Minimum erythema dose (MED)baseline to MEDon-drug at each respective post irradiation time point (i.e. 1 hour)(i.e., MEDon-drug[millijoules (mJ)]/MEDbaseline[mJ]) and was hence unitless.
  MED was defined as lowest dose that produced uniform redness (C1) (assessed in mJ for UVB/UVA).
  Subjects were exposed to a series of 6 graded full range solar UVB/UVA exposures, each 25% greater than the previous dose.
  Light exposure occurred 2 hours (±10 minutes) after dose on Day 8 of either investigational product (IP) or placebo, and on-treatment photosensitivity assessments (determination of MEDon-drug + evaluation of erythema/local skin reactions) were performed at 1 hour after irradiation.
Time Frame: At 1 hour after irradiation on Day 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Unitless
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Number analyzed (Participants) | 8 | 27 | 7 | 25 | 12
Unitless | 1.07 [0.99 to 1.15] | 0.99 [0.95 to 1.03] | 1.04 [0.85 to 1.22] | 1.08 [0.99 to 1.18] | 1.00 [0.94 to 1.06]
Statistical Analysis 1: Comparison: Placebo QD vs 400 mg QD BI 730357; Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; Test type: Equivalence — Two-sided 90% CI with an acceptance range of -0.4 to 0.4; Linear mixed model; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.08, 90% CI 2-sided [-0.15 to -0.01], Standard Error of Mean 0.043
Statistical Analysis 2: Comparison: 400 mg QD BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.757, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.01, 90% CI 2-sided [-0.09 to 0.06], Standard Error of Mean 0.037
Statistical Analysis 3: Comparison: Placebo QD vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.158, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.07, 90% CI 2-sided [-0.17 to 0.03], Standard Error of Mean 0.049
Statistical Analysis 4: Comparison: Placebo BID vs 300 mg BID BI 730357; Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; Test type: Equivalence — Two-sided 90% CI with an acceptance range of -0.4 to 0.4; Linear mixed model; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.05, 90% CI 2-sided [-0.12 to 0.22], Standard Error of Mean 0.101
Statistical Analysis 5: Comparison: 300 mg BID BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.330, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.08, 90% CI 2-sided [-0.09 to 0.25], Standard Error of Mean 0.083
Statistical Analysis 6: Comparison: Placebo BID vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.754, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.04, 90% CI 2-sided [-0.26 to 0.19], Standard Error of Mean 0.113

6. Secondary Outcome: Photosensitivity Index (PI) at 1 Hour Under Condition 2 (i.e., Under UVA Exposure Only, Simulating Indoor Sun Exposure Behind Window Glass)
Description: Photosensitivity index (PI) under condition 2 (C2)(i.e., UVA only (320 to 400 nm, UVB content <0.03%), simulating indoor exposure behind window glass with a secondary assessment of erythema and local skin reactions at 25 Joules centimetres-2 (J cm-2) (assessed in mw/cm2)), defined as ratio of precise Minimum erythema dose (MED)baseline to MEDon-drug at each respective post irradiation time point (i.e. 1 hour)(i.e. MEDon-drug[Joules (J)]/MEDbaseline[J]) and was hence unitless.
  MED defined as lowest dose that produced uniform darkening (C2) (assessed in J for UVA).
  Subjects were exposed to series of 6 graded full range solar UVA only exposures (C2), each 25% greater than the previous dose.
  Light exposure occurred 2 hours (±10 minutes) after dose on Day 8 of either investigational product (IP) or placebo, and on-treatment photosensitivity assessments (determination of MEDon-drug + evaluation of erythema/local skin reactions) were performed at 1 hour after irradiation.
Time Frame: At 1 hour after irradiation on Day 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Unitless
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Number analyzed (Participants) | 8 | 27 | 7 | 25 | 12
Unitless | 0.91 [0.68 to 1.14] | 1.22 [1.10 to 1.34] | 1.00 [0.76 to 1.24] | 1.19 [1.06 to 1.32] | 1.06 [0.87 to 1.24]
Statistical Analysis 1: Comparison: Placebo QD vs 400 mg QD BI 730357; Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; Test type: Equivalence — Two-sided 90% CI with an acceptance range of -0.4 to 0.4; Linear mixed model; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.31, 90% CI 2-sided [0.09 to 0.52], Standard Error of Mean 0.128
Statistical Analysis 2: Comparison: 400 mg QD BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.151, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.16, 90% CI 2-sided [-0.06 to 0.38], Standard Error of Mean 0.110
Statistical Analysis 3: Comparison: Placebo QD vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.319, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.15, 90% CI 2-sided [-0.15 to 0.44], Standard Error of Mean 0.145
Statistical Analysis 4: Comparison: Placebo BID vs 300 mg BID BI 730357; Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; Test type: Equivalence — Two-sided 90% CI with an acceptance range of -0.4 to 0.4; Linear mixed model; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.19, 90% CI 2-sided [-0.04 to 0.42], Standard Error of Mean 0.136
Statistical Analysis 5: Comparison: 300 mg BID BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.246, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.13, 90% CI 2-sided [-0.09 to 0.36], Standard Error of Mean 0.112
Statistical Analysis 6: Comparison: Placebo BID vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.704, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.06, 90% CI 2-sided [-0.25 to 0.36], Standard Error of Mean 0.151

7. Secondary Outcome: Minimum Erythema Dose (MED) Percent Change From Baseline at 10 Minutes Under Condition 1 (i.e., Under Full Range of UVB/UVA Exposure, Simulating Midday Summer Outdoor Sun Exposure)
Description: The Minimum erythema dose (MED) percent change from baseline at 10 minutes was calculated as follows: % change = ([MEDon-drug - MEDbaseline]/ MEDbaseline) x 100.
  MED under condition 1 (C1)(i.e., under full range solar UVB/UVA (290 to 400 nm, UBV content ~10%), simulating midday summer outdoor sun exposure (assessed in μw/cm2)), was defined as lowest dose that produced uniform redness (assessed in mJ for UVB/UVA).
  Subjects were exposed to a series of 6 graded full range solar UVB/UVA exposures, each 25% greater than the previous dose.
  Light exposure occurred 2 hours (±10 minutes) after dose on Day 8 of either investigational product (IP) or placebo, and on-treatment photosensitivity assessments (determination of MEDon-drug + evaluation of erythema/local skin reactions) were performed at 10 minutes after irradiation.
Time Frame: At baseline (Day -2) and at 10 minutes after irradiation on Day 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Number analyzed (Participants) | 8 | 27 | 7 | 25 | 12
Percent change | 3.12 [-4.88 to 11.12] | 1.68 [-2.68 to 6.03] | 0.00 [-8.80 to 8.80] | -1.96 [-6.62 to 2.69] | 0.00 [-6.53 to 6.53]
Statistical Analysis 1: Comparison: Placebo BID vs 300 mg BID BI 730357; Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.692, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -1.96, 90% CI 2-sided [-11.92 to 7.99], Standard Error of Mean 4.929
Statistical Analysis 2: Comparison: 300 mg BID BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.630, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -1.96, 90% CI 2-sided [-10.14 to 6.21], Standard Error of Mean 4.048
Statistical Analysis 3: Comparison: Placebo BID vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 1.000, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.00, 90% CI 2-sided [-11.07 to 11.07], Standard Error of Mean 5.482
Statistical Analysis 4: Comparison: Placebo QD vs 400 mg QD BI 730357; Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.751, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -1.44, 90% CI 2-sided [-10.55 to 7.66], Standard Error of Mean 4.518
Statistical Analysis 5: Comparison: 400 mg QD BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.669, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 1.68, 90% CI 2-sided [-6.17 to 9.52], Standard Error of Mean 3.894
Statistical Analysis 6: Comparison: Placebo QD vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.546, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -3.12, 90% CI 2-sided [-13.44 to 7.21], Standard Error of Mean 5.123

8. Secondary Outcome: Minimum Erythema Dose (MED) Percent Change From Baseline at 10 Minutes Under Condition 2 (i.e., Under UVA Exposure Only, Simulating Indoor Sun Exposure Behind Window Glass)
Description: The Minimum erythema dose (MED) percent change from baseline at 10 minutes was calculated as follows: % change = ([MEDon-drug - MEDbaseline]/ MEDbaseline) x 100.
  MED under condition 2 (C2)(i.e., UVA only (320 to 400 nm, UVB content <0.03%), simulating indoor exposure behind window glass with a secondary assessment of erythema and local skin reactions at 25 Joules centimetres-2 (J cm-2) (assessed in mw/cm2)), was defined as lowest dose that produced uniform darkening (assessed in J for UVA).
  Subjects were exposed to a series of 6 graded full range solar UVA only exposures, each 25% greater than the previous dose.
  Light exposure occurred 2 hours (±10 minutes) after dose on Day 8 of either investigational product (IP) or placebo, and on-treatment photosensitivity assessments (determination of MEDon-drug + evaluation of erythema/local skin reactions) were performed at 10 minutes after irradiation.
Time Frame: At baseline (Day -2) and at 10 minutes after irradiation on Day 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Number analyzed (Participants) | 8 | 27 | 7 | 25 | 12
Percent change | 7.19 [-16.27 to 30.66] | -1.02 [-13.79 to 11.75] | 0.00 [-20.32 to 20.32] | -12.45 [-23.20 to -1.69] | 3.69 [-15.46 to 22.85]
Statistical Analysis 1: Comparison: Placebo BID vs 300 mg BID BI 730357; Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.281, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -12.45, 90% CI 2-sided [-35.44 to 10.54], Standard Error of Mean 11.385
Statistical Analysis 2: Comparison: 300 mg BID BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.092, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -16.14, 90% CI 2-sided [-35.02 to 2.74], Standard Error of Mean 9.350
Statistical Analysis 3: Comparison: Placebo BID vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.772, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 3.69, 90% CI 2-sided [-21.88 to 29.27], Standard Error of Mean 12.662
Statistical Analysis 4: Comparison: Placebo QD vs 400 mg QD BI 730357; Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.539, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -8.21, 90% CI 2-sided [-34.93 to 18.50], Standard Error of Mean 13.255
Statistical Analysis 5: Comparison: 400 mg QD BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.682, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -4.71, 90% CI 2-sided [-27.74 to 18.31], Standard Error of Mean 11.424
Statistical Analysis 6: Comparison: Placebo QD vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.817, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -3.50, 90% CI 2-sided [-33.79 to 26.79], Standard Error of Mean 15.030

9. Secondary Outcome: Minimum Erythema Dose (MED) Percent Change From Baseline at 1 Hour Under Condition 1 (i.e., Under Full Range of UVB/UVA Exposure, Simulating Midday Summer Outdoor Sun Exposure)
Description: The Minimum erythema dose (MED) percent change from baseline at 1 hour was calculated as follows: % change = ([MEDon-drug - MEDbaseline]/ MEDbaseline) x 100.
  MED under condition 1 (C1)(i.e., under full range solar UVB/UVA (290 to 400 nm, UBV content ~10%), simulating midday summer outdoor sun exposure (assessed in μw/cm2)), was defined as lowest dose that produced uniform redness (assessed in mJ for UVB/UVA).
  Subjects were exposed to a series of 6 graded full range solar UVB/UVA exposures, each 25% greater than the previous dose.
  Light exposure occurred 2 hours (±10 minutes) after dose on Day 8 of either investigational product (IP) or placebo, and on-treatment photosensitivity assessments (determination of MEDon-drug + evaluation of erythema/local skin reactions) were performed at 1 hour after irradiation.
Time Frame: At baseline (Day -2) and at 1 hour after irradiation on Day 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Number analyzed (Participants) | 8 | 27 | 7 | 25 | 12
Percent change | -4.50 [-12.26 to 3.26] | 2.29 [-1.94 to 6.51] | -2.85 [-12.36 to 6.66] | -3.59 [-8.62 to 1.44] | 0.00 [-7.26 to 7.26]
Statistical Analysis 1: Comparison: Placebo BID vs 300 mg BID BI 730357; Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.891, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -0.73, 90% CI 2-sided [-11.49 to 10.02], Standard Error of Mean 5.327
Statistical Analysis 2: Comparison: 300 mg BID BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.417, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -3.59, 90% CI 2-sided [-12.42 to 5.25], Standard Error of Mean 4.375
Statistical Analysis 3: Comparison: Placebo BID vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.633, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 2.85, 90% CI 2-sided [-9.11 to 14.82], Standard Error of Mean 5.925
Statistical Analysis 4: Comparison: Placebo QD vs 400 mg QD BI 730357; Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.129, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 6.79, 90% CI 2-sided [-2.05 to 15.62], Standard Error of Mean 4.384
Statistical Analysis 5: Comparison: 400 mg QD BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.548, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 2.29, 90% CI 2-sided [-5.33 to 9.90], Standard Error of Mean 3.778
Statistical Analysis 6: Comparison: Placebo QD vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.370, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 4.50, 90% CI 2-sided [-5.51 to 14.52], Standard Error of Mean 4.970

10. Secondary Outcome: Minimum Erythema Dose (MED) Percent Change From Baseline at 1 Hour Under Condition 2 (i.e., Under UVA Exposure Only, Simulating Indoor Sun Exposure Behind Window Glass)
Description: The Minimum erythema dose (MED) percent change from baseline at 1 hour was calculated as follows: % change = ([MEDon-drug - MEDbaseline]/ MEDbaseline) x 100.
  MED under condition 2 (C2)(i.e., UVA only (320 to 400 nm, UVB content <0.03%), simulating indoor exposure behind window glass with a secondary assessment of erythema and local skin reactions at 25 Joules centimetres-2 (J cm-2) (assessed in mw/cm2)), was defined as lowest dose that produced uniform darkening (assessed in J for UVA).
  Subjects were exposed to a series of 6 graded full range solar UVA only exposures, each 25% greater than the previous dose.
  Light exposure occurred 2 hours (±10 minutes) after dose on Day 8 of either investigational product (IP) or placebo, and on-treatment photosensitivity assessments (determination of MEDon-drug + evaluation of erythema/local skin reactions) were performed at 1 hour after irradiation.
Time Frame: At baseline (Day -2) and at 1 hour after irradiation on Day 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Number analyzed (Participants) | 8 | 27 | 7 | 25 | 12
Percent change | 13.82 [-2.83 to 30.47] | -12.82 [-21.88 to -3.76] | 0.00 [-18.53 to 18.53] | -9.30 [-19.10 to 0.50] | 2.19 [-11.40 to 15.78]
Statistical Analysis 1: Comparison: Placebo BID vs 300 mg BID BI 730357; Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.375, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -9.30, 90% CI 2-sided [-30.26 to 11.66], Standard Error of Mean 10.379
Statistical Analysis 2: Comparison: 300 mg BID BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.185, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -11.49, 90% CI 2-sided [-28.70 to 5.73], Standard Error of Mean 8.524
Statistical Analysis 3: Comparison: Placebo BID vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.851, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 2.19, 90% CI 2-sided [-21.12 to 25.50], Standard Error of Mean 11.544
Statistical Analysis 4: Comparison: Placebo QD vs 400 mg QD BI 730357; Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.007, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -26.64, 90% CI 2-sided [-45.59 to -7.69], Standard Error of Mean 9.405
Statistical Analysis 5: Comparison: 400 mg QD BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.071, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -15.01, 90% CI 2-sided [-31.34 to 1.33], Standard Error of Mean 8.106
Statistical Analysis 6: Comparison: Placebo QD vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.281, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -11.63, 90% CI 2-sided [-33.13 to 9.86], Standard Error of Mean 10.664

11. Secondary Outcome: Minimum Erythema Dose (MED) Percent Change From Baseline at 24 Hours Under Condition 1 (i.e., Under Full Range of UVB/UVA Exposure, Simulating Midday Summer Outdoor Sun Exposure)
Description: The Minimum erythema dose (MED) percent change from baseline at 24 hours was calculated as follows: % change = ([MEDon-drug - MEDbaseline]/ MEDbaseline) x 100.
  MED under condition 1 (C1)(i.e., under full range solar UVB/UVA (290 to 400 nm, UBV content ~10%), simulating midday summer outdoor sun exposure (assessed in μw/cm2)), was defined as lowest dose that produced uniform redness (assessed in mJ for UVB/UVA).
  Subjects were exposed to a series of 6 graded full range solar UVB/UVA exposures, each 25% greater than the previous dose.
  Light exposure occurred 2 hours (±10 minutes) after dose on Day 8 of either investigational product (IP) or placebo, and on-treatment photosensitivity assessments (determination of MEDon-drug + evaluation of erythema/local skin reactions) were performed at 24 hours after irradiation.
Time Frame: At baseline (Day -2) and at 24 hours after irradiation on Day 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Number analyzed (Participants) | 8 | 27 | 7 | 25 | 12
Percent change | 9.35 [-2.80 to 21.51] | 1.35 [-5.26 to 7.97] | 0.00 [-9.59 to 9.59] | -2.84 [-7.92 to 2.23] | -3.83 [-11.15 to 3.49]
Statistical Analysis 1: Comparison: Placebo BID vs 300 mg BID BI 730357; Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.599, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -2.84, 90% CI 2-sided [-13.69 to 8.00], Standard Error of Mean 5.370
Statistical Analysis 2: Comparison: 300 mg BID BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.824, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.99, 90% CI 2-sided [-7.92 to 9.90], Standard Error of Mean 4.410
Statistical Analysis 3: Comparison: Placebo BID vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.525, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -3.83, 90% CI 2-sided [-15.90 to 8.23], Standard Error of Mean 5.973
Statistical Analysis 4: Comparison: Placebo QD vs 400 mg QD BI 730357; Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.250, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -8.00, 90% CI 2-sided [-21.84 to 5.84], Standard Error of Mean 6.867
Statistical Analysis 5: Comparison: 400 mg QD BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.386, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 5.19, 90% CI 2-sided [-6.74 to 17.12], Standard Error of Mean 5.919
Statistical Analysis 6: Comparison: Placebo QD vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.097, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -13.19, 90% CI 2-sided [-28.88 to 2.51], Standard Error of Mean 7.787

12. Secondary Outcome: Minimum Erythema Dose (MED) Percent Change From Baseline at 24 Hours Under Condition 2 (i.e., Under UVA Exposure Only, Simulating Indoor Sun Exposure Behind Window Glass)
Description: The Minimum erythema dose (MED) percent change from baseline at 24 hours was calculated as follows: % change = ([MEDon-drug - MEDbaseline]/ MEDbaseline) x 100.
  MED under condition 2 (C2)(i.e., UVA only (320 to 400 nm, UVB content <0.03%), simulating indoor exposure behind window glass with a secondary assessment of erythema and local skin reactions at 25 Joules centimetres-2 (J cm-2) (assessed in mw/cm2)), was defined as lowest dose that produced uniform darkening (assessed in J for UVA).
  Subjects were exposed to a series of 6 graded full range solar UVA only exposures, each 25% greater than the previous dose.
  Light exposure occurred 2 hours (±10 minutes) after dose on Day 8 of either investigational product (IP) or placebo, and on-treatment photosensitivity assessments (determination of MEDon-drug + evaluation of erythema/local skin reactions) were performed at 24 hours after irradiation.
Time Frame: At baseline and at 24 hours
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo QD | 400 mg QD BI 730357 | Placebo BID | 300 mg BID BI 730357 | 500 mg Ciprofloxacin (Active Comparator)
Number analyzed (Participants) | 8 | 27 | 7 | 25 | 12
Percent change | 10.71 [-3.52 to 24.95] | -9.41 [-17.16 to -1.67] | 0.00 [-12.21 to 12.21] | 0.99 [-5.47 to 7.46] | -27.91 [-39.53 to -16.29]
Statistical Analysis 1: Comparison: Placebo BID vs 300 mg BID BI 730357; Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.885, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 0.99, 90% CI 2-sided [-12.83 to 14.81], Standard Error of Mean 6.842
Statistical Analysis 2: Comparison: 300 mg BID BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p < 0.001, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 28.90, 90% CI 2-sided [17.55 to 40.25], Standard Error of Mean 5.619
Statistical Analysis 3: Comparison: Placebo BID vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p < 0.001, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -27.91, 90% CI 2-sided [-43.28 to -12.54], Standard Error of Mean 7.610
Statistical Analysis 4: Comparison: Placebo QD vs 400 mg QD BI 730357; Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.016, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -20.13, 90% CI 2-sided [-36.33 to -3.92], Standard Error of Mean 8.041
Statistical Analysis 5: Comparison: 400 mg QD BI 730357 vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p = 0.011, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = 18.50, 90% CI 2-sided [4.53 to 32.46], Standard Error of Mean 6.931
Statistical Analysis 6: Comparison: Placebo QD vs 500 mg Ciprofloxacin (Active Comparator); Test type: Other — Mixed model for repeated measures (MMRM) with unstructured (UN) covariance matrix on photosensitivity index (PI) values; p < 0.001, Linear mixed model — P-value is for testing Least Squares Mean Difference=0; Treatment, time, and treatment-time interaction as fixed effects and subject as a random effect; Mean Difference (Final Values) = -38.62, 90% CI 2-sided [-57.00 to -20.25], Standard Error of Mean 9.118

ADVERSE EVENTS:
Time Frame: From start of treatment until end of the 7 day follow up period, 15 days in total.
Description: Treated Set (TS): The TS included all subjects who were randomized and treated with at least 1 dose of investigational product (IP) (BI 730357, placebo, or Ciprofloxacin). The TS was used for safety analyses.
Groups:
- Placebo QD/BID: Subjects received orally, four Placebo film-coated tablets once per day (QD) over 8 days or three Placebo film-coated tablets two times per day (BID) over 7 days with a single dose on Day 8. Medication administration was to take place at the same time every day within a deviation of no more than ±15 minutes together with about 240 mL of water.
- 500 mg BID Ciprofloxacin (Active Comparator)): Subjects received orally, one Ciprofloxacin film-coated tablet of 500 miligrams (mg) each, two times per days (BID) (2 x 500 mg = 1000 mg in total) over 5 days from day 3 with a single dose on Day 8. Medication administration was to take place at the same time every day within a deviation of no more than ±15 minutes together with about 240 mL of water.
Arm/Group | Placebo QD/BID | 400 mg QD BI 730357 | 300 mg BID BI 730357 | 500 mg BID Ciprofloxacin (Active Comparator))
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/27 | 0/28 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/27 | 0/28 | 0/12
Other Adverse Events (participants affected / at risk) | 7/18 | 9/27 | 11/28 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD/BID (N=18) | 400 mg QD BI 730357 (N=27) | 300 mg BID BI 730357 (N=28) | 500 mg BID Ciprofloxacin (Active Comparator)) (N=12)
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 5 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 4 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 3 | 0
Headache (Nervous system disorders) | 3 | 6 | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT04147260/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT04147260/SAP_001.pdf